CLINICAL TRIAL: NCT02092857
Title: Assessment of Arachidonic Acid Supplementation in Infant Formula on the Immune Response of Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00005583; 230831 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Focus: Nutritional Requirements for Infants
Keywords: nutrient; nutrition; arachidonic acid; essential fatty acids
MeSH Terms: interventions — Arachidonic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 34 mg/100 kcal arachidonic acid (Active Comparator): 10 weeks exclusive feeding with infant formula containing 34 mg/100 kcal of arachidonic acid
  Interventions: Dietary Supplement: Arachidonic acid (34 mg/100 kcal)
- 25 mg/100 kcal arachidonic acid (Active Comparator): 10 weeks exclusive feeding with infant formula containing 25 mg/100 kcal of arachidonic acid
  Interventions: Dietary Supplement: Arachidonic acid (25 mg/100 kcal )
- Infant formula without arachidonic acid (Placebo Comparator): 10 weeks exclusive infant formula feeding (without supplemental arachidonic acid).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Arachidonic acid (25 mg/100 kcal )
  Arms: 25 mg/100 kcal arachidonic acid
Dietary Supplement: Arachidonic acid (34 mg/100 kcal)
  Arms: 34 mg/100 kcal arachidonic acid
Dietary Supplement: Placebo — 10 weeks exclusive infant formula feeding (without supplemental arachidonic acid).
  Arms: Infant formula without arachidonic acid

SUMMARY:
The immune system of newborn infants is immature with low activity of both innate and acquired immune reactions. Early nutrition has an impact on early immune responses. Dietary fatty acids are one nutritional factor noted to play a role in immune function. The omega-6 long-chain polyunsaturated fatty acid, ARA (Arachidonic acid) and the omega-3 fatty acid, DHA (docosahexaenoic acid) are found naturally in breastmilk and some infant formulas. The balance or relative amounts of ARA and DHA have been associated with immune response. Some commercial infant formula contains both ARA and DHA. However, the optimal balance of ARA and DHA has not been determined with respect to immune function. This study will assess two levels of ARA and the impact on immune response in healthy, term infants and whether genes that influence essential fatty acid metabolism alter the nutritional requirement of infants.

ELIGIBILITY:
Inclusion criteria:

* healthy term infants
* birth weight, length and head circumference between the 5th and 95th percentile for gestational age (according to the National Center for Health Statistics growth charts)
* receiving >80% for their intake by mouth from commercial infant formula
* low-risk for allergy based on a negative family history.

Exclusion criteria:

* corticosteroid use
* red cell or plasma transfusions
* IV lipid emulsions prior to study entry
* major congenital malformations
* systemic or congenital infection
* significant neonatal morbidity
* maternal autoimmune disorders
* acute illness precluding oral feedings or conditions requiring feedings other than standard formula

Ages: 14 Days to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Clandinin, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 34 mg/100 kcal Arachidonic Acid | 25 mg/100 kcal Arachidonic Acid | Infant Formula Without Arachidonic Acid
Started | 30 | 30 | 29
Completed | 20 | 18 | 16
Not Completed | 10 | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 34 mg/100 kcal Arachidonic Acid | 25 mg/100 kcal Arachidonic Acid | Infant Formula Without Arachidonic Acid | Total
Number analyzed (Participants) | 30 | 30 | 29 | 89
Age, Continuous [Mean (Standard Deviation); unit: days] | 16.8 (3.8) | 16.5 (3.8) | 17.8 (4.4) | 17 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 16 | 48
  Male | 15 | 13 | 13 | 41
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 30 | 29 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Antigen-presenting B Cells
Time Frame: 10 weeks
Measure: Number; unit: percentage of CD20+ B cells
Arm/Group | 34 mg/100 kcal Arachidonic Acid | 25 mg/100 kcal Arachidonic Acid | Infant Formula Without Arachidonic Acid
Number analyzed (Participants) | 13 | 12 | 9
percentage of CD20+ B cells | 21.9 | 22.8 | 25.1

ADVERSE EVENTS:
Arm/Group | 34 mg/100 kcal Arachidonic Acid | 25 mg/100 kcal Arachidonic Acid | Infant Formula Without Arachidonic Acid
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 2/30 | 7/30 | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 34 mg/100 kcal Arachidonic Acid (N=30) | 25 mg/100 kcal Arachidonic Acid (N=30) | Infant Formula Without Arachidonic Acid (N=29)
sudden unexpected infant death (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 34 mg/100 kcal Arachidonic Acid (N=30) | 25 mg/100 kcal Arachidonic Acid (N=30) | Infant Formula Without Arachidonic Acid (N=29)
swallowing disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
gastroesophageal reflux (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
colic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
cow's milk intolerance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
inguinal hernia - male (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes